CLINICAL TRIAL: NCT03057002
Title: Detection of Myocardial Metabolic Changes in Patients With Cardiomyopathy Using Hyperpolarized Carbon 13 Magnetic Resonance Spectroscopic Imaging
Brief Title: UTSW HP [13-C] Pyruvate Injection in HCM
Acronym: HPHCM
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vlad Zaha, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 102016-046
Record Dates: First submitted 2017-01-10; First posted 2017-02-17 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathy, Hypertrophic; Dilated Cardiomyopathy; Duchenne Muscular Dystrophy; Cardiac Sarcoidosis; Becker Muscular Dystrophy; Heart Failure With Preserved Ejection Fraction; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cardiomyopathy: Patients with Cardiomyopathy will be observed for myocardial hyperpolarized 13C-pyruvate flux during magnetic resonance spectroscopic imaging.
  Interventions: Diagnostic Test: Hyperpolarized 13C-Pyruvate
- Control: Healthy control subjects will be observed for myocardial hyperpolarized 13C-pyruvate flux during magnetic resonance spectroscopic imaging.
  Interventions: Diagnostic Test: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Diagnostic Test: Hyperpolarized 13C-Pyruvate — All subjects will be observed for myocardial hyperpolarized [1-13C]pyruvate flux during magnetic resonance spectroscopic imaging.
  Other Names: HP [1-13C]pyruvate

SUMMARY:
The study objective is to identify the earliest changes in energy substrate metabolism in patients with cardiomyopathies (CMP). To achieve this objective, we plan first to test the hypothesis that patients with CMP present focal alterations in myocardial hyperpolarized [1-13C]pyruvate flux.

DETAILED DESCRIPTION:
To measure the regional myocardial [1-13C]lactate to [13C]bicarbonate ratio as an index of mitochondrial oxidation and glycolysis coupling in the heart. Advanced cardiac MRI will be used to characterize cardiac morphology, function, myocardial blood flow and fibrosis.

Heart failure is a major source of morbidity and mortality in the United States. Multiple studies have demonstrated that development of heart failure is related to alteration in cardiac metabolism. Specifically, such changes include a shift from fatty acid oxidation to increased glucose utilization as energy source, with uncoupling of glycolysis and mitochondrial oxidation at the level of the pyruvate dehydrogenase complex. In human subject who were referred for LVAD placement, excised heart muscle samples exhibited significant increase in expression of pyruvate kinase M2 (PKM2) compared to subjects with normal LV function.

Additionally, mechanical unloading decreased PKM2 expression suggesting a correlation between pyruvate utilization and severity of heart failure. Such changes metabolic alterations appear to precede the actual structural changes and might be a possible target for future therapies, although the timeline of such changes remains to be elucidated. Currently, it is unknown whether different types of CMP have different metabolic signatures.

ELIGIBILITY:
Inclusion Criteria for Control Subjects:

* Subjects who are 18.
* Subjects who have the ability to understand and the willingness to sign a written informed consent.
* While all races and ethnicities will be included, subjects must be able to read and speak the English language. Once the protocol is established, Spanish-speaking participants will be included.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Inclusion Criteria for participants with Cardiomyopathy:

* Subjects who are 18.
* Subjects who have the ability to understand and the willingness to sign a written informed consent.
* While all races and ethnicities will be included, subjects must be able to read and speak the English language. Once the protocol is established, Spanish-speaking participants will be included.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion criteria:

* Subjects who are receiving any other investigational agents.
* Intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled chronic diseases such as hypertension, lung disease, liver disease, kidney disease, diabetes, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects who are taking thyroid hormone replacements, have a history of alcohol abuse or illicit drug use.
* Subjects who have contraindication to contrast enhanced MRI examination.

Contraindications to MRI examinations include:

* Medically unstable
* Acute Heart failure
* Severe LVOT obstruction
* Unstable angina
* Child bearing
* Lactating
* Any contraindication per MRI Screening Form including
* Implants contraindicated at 3Tesla, pacemakers
* Implantable Cardioverter Defibrillator (ICD)
* Claustrophobia
* Since each subject is receiving a gadolinium based contrast agent intravenously:
* eGFR ≤ 30 mL/min/1.73m2
* Sickle cell disease
* Hemolytic anemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 5 Cardiomyopathy (CMP) Patients and 5 Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Hyperpolarized [1-13C]pyruvate flux | Screening (Baseline) and 1 day of Study Visit
  Measurement of change in myocardial hyperpolarized [1-13C]pyruvate flux during Magnetic Resonance Spectroscopic Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Vlad G Zaha, MD, PhD, Principal Investigator — Advanced Imaging Research Center
Locations (1):
- UT Southwestern Medical Center - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No